CLINICAL TRIAL: NCT02933593
Title: Changes in Central Arterial Pressure When Comparing ACOG Hypertensive Urgency Protocols
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI withdrew the protocol
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Jennifer Goldkamp, MD, Principal Investigator, St. Louis University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 27295
Record Dates: First submitted 2016-08-22; First posted 2016-10-14 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Labetalol; Hydralazine; Nifedipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- labetalol (Active Comparator): labetalol
  Interventions: Drug: Labetalol
- hydralazine (Active Comparator): Hydralazine
  Interventions: Drug: Hydralazine
- nifedipine (Active Comparator): nifedipine
  Interventions: Drug: nifedipine

INTERVENTIONS:
Drug: Labetalol — To determine which protocol recommended by ACOG for severe hypertension in pregnancy decreases central arterial pressure the fastest, and the most efficaciously.
  Other Names: Trandate®
  Arms: labetalol
Drug: Hydralazine — To determine which protocol recommended by ACOG for severe hypertension in pregnancy decreases central arterial pressure the fastest, and the most efficaciously.
  Other Names: Apresoline
  Arms: hydralazine
Drug: nifedipine — To determine which protocol recommended by ACOG for severe hypertension in pregnancy decreases central arterial pressure the fastest, and the most efficaciously.
  Other Names: Procardia
  Arms: nifedipine

SUMMARY:
The investigators plan to monitor the central blood pressure in women with severely elevated blood pressures (160/110) in pregnancy in the acute setting. Currently ACOG recommends 3 different options for blood pressure control, however no one has studied how these medications affect the central pressures, only peripheral blood pressure.

DETAILED DESCRIPTION:
Women will be screened as they come in through the Women's Evaluation Unit or as transfers from outside hospitals to Labor & Delivery or the Perinatal Special Care Unit (PSCU). All women with severe hypertension (defined as 160/110 or above for 15 minutes or more) will be screened for inclusion and asked to participate in the study. If the woman agrees to participate she will be randomized to one of three groups with the following protocol:

Labetalol Administer 20mg IV labetalol Repeat BP in 10 minutes, if still severe administer 40mg IV Labetalol Repeat BP in 10 minutes, if still elevated administer 80mg IV Labetalol Repeat BP in 10 minutes, if still elevated administer 10mg IV Hydralazine Repeat BP in 20 minutes, if still elevated consider ICU consult Hydralazine Administer 5mg IV hydralazine Repeat BP in 20 minutes, if still elevated administer 10mg IV Hydralazine Repeat BP in 20 minutes, still elevated administer labetalol 20mg IV Repeat BP in 10 minutes, still elevated administer labetalol 40mg IV and consider ICU consult Nifedipine Administer procardia 10mg po Repeat BP in 20 min, if still elevated administer procardia 20mg po Repeat BP in 20 min, if still elevated administer procardia 20mg po Repeat BP in 20 min, if still elevated administer labetalol 40mg IV and consider ICU consult

Administration of medication will be determined by the routine sphygmomanometer blood pressure as that is what the guidelines are based upon.

Women will then have their central arterial pressure and their carotid waveform assessed before administration of medication. The central pressure will be assessed every 5 minutes and carotid waveforms every 10 minutes until blood pressures are <160/110 for 20 minutes.

Administration of the above medications is standard of care. Randomization to different medications, measuring the central pressure and the carotid waveform is part of the study.

Once the patient's BP stays below 160/110 for 20 minutes their participation in the study will end.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Singleton pregnancy
* Severe hypertension as defined by a blood pressure of 160/110 with plans to treat

Exclusion Criteria:

* Multiple pregnancy
* Blood pressures < 160/110, or those whose blood pressures do not require medication for control
* Irregular heart rhythms or arrhythmias
* Peripheral arterial disease, leg artery disease
* Reynaud's phenomena
* Intense cold/hypothermia
* If there is a wound at location of where central arterial cuff would be placed or tonometer for carotid assessment
* Known sensitivity to labetalol, nifedipine, or hydralazine
* Severe tachycardia (>120)
* Greater than 1st degree heart block
* Severe asthma
* Congestive heart failure or heart disease
* Lupus
* Inability to adequately monitor BP
* Inability to monitor fetus (if 23 weeks or above)
* Magnesium started prior to initiation of study

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
medication recommended by ACOG for severe hypertension | 20min from time of first normal blood pressure after intervention
  To determine which protocol recommended by ACOG for severe hypertension in pregnancy decreases central arterial pressure the fastest, and the most efficaciously

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Goldkamp, MD, Principal Investigator — St. Louis University

IPD SHARING:
Plan to Share IPD: No